CLINICAL TRIAL: NCT04792008
Title: A Randomised, Double-Blind, Phase 1b/2a, Placebo-Controlled, Single Dose Study to Evaluate Safety, Tolerability, and Efficacy of YQ23 in Adult Patients With Critical Limb Ischaemia
Brief Title: YQ23 Study in Patients With Critical Limb Ischaemia
Acronym: YAN
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to business decision
Sponsor: New Beta Innovation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YQ23-19001
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-03

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YQ23 Single dose (Experimental): Two-third of randomized patients will receive YQ23 as active treatment
  Interventions: Biological: YQ23
- Placebo Single dose (Placebo Comparator): One-third of randomized patients will receive matching placebo
  Interventions: Biological: Matching placebo

INTERVENTIONS:
Biological: YQ23 — Single dose of 120 mg/kg YQ23 via intravenous route will be evaluated
  Arms: YQ23 Single dose
Biological: Matching placebo — Single dose of 0.9% normal saline via intravenous route as matching placebo
  Arms: Placebo Single dose

SUMMARY:
This is an early phase study to assess how safe and tolerable is the new study drug YQ23 and to compare the effectiveness of YQ23 against normal saline to treat critical limb ischaemia. The study also aims to understand how it affects the body and an optional substudy to assess how the human body takes up, breaks down, and clears the study drug.

Eligible patients will be randomised to have a 2:1 chance to receive a single, intravenous, fixed dose of YQ23 or normal saline. Neither the patient nor the study site will know which treatment has been given.

On the day of YQ23 administration, patients will be asked to stay in the study site for 3 days for safety observation. After discharge, they will be required to visit the study clinic for 3 times in a year to continue safety monitoring and assessment of treatment effect.

Each subject's participation will be about 13 months after signing the informed consent.

DETAILED DESCRIPTION:
This is a Phase 1b/2a, randomised, double-blind, placebo-controlled study to evaluate the safety, tolerability, and efficacy of an investigational product, YQ23, in patients with Critical Limb Ischaemia (CLI) during a follow-up period of 12 months.

Fifty-one patients are planned for enrolment. The study consists of a screening period (up to 28 days), a double-blind treatment period, and a follow-up (12 months). Prior to randomisation, patients diagnosed with CLI will be stratified into:

* Group of patients in whom revascularisation is not planned
* Group of patients with planned revascularisation

Within each group, patients will be randomised in a 2:1 ratio to receive single intravenous infusion of YQ23 120 mg/kg and normal saline, respectively at the study site.

On the day of YQ23 administration, the patient will be admitted to the study site on Day 1 and will be discharged on Day 3. The total duration of participation in the study for each patient is approximately 13 months. Data on the study endpoints will be collected from baseline (pre-dose on Day 1), Day 3, Month 1, 6 and up to 12 months after study treatment infusion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLI (Rutherford Classification stage 4, 5 or 6) including at least one of the following:

  1. resting ankle systolic pressure (either dorsalis pedis or posterior tibial artery) <=70 mmHg in affected limb
  2. resting toe systolic pressure <=50 mmHg in affected limb
  3. TcPO2 <=30 mmHg
* One of the following clinical presentations:

  1. pain at rest
  2. ischaemic ulcer, and/or focal gangrene for at least 2 weeks
* Diagnosis of severe lower extremity peripheral artery occlusive disease as evidenced by either:

  1. Documented significant stenosis (>=75%) of >=1 of the following arteries: superficial femoral, popliteal, and infra-popliteal arteries, as assessed by imaging test, or
  2. ABI <=0.80 or TBI <=0.60 of the index leg (in the event of non-compressible ankle arteries) for patients without a prior history of limb revascularization on the index leg, or an ABI <=0.85 or TBI <=0.65 of the index leg (in the event of non-compressible ankle arteries) for patients with a prior history of limb revascularization on the index leg.
* Contraceptive use

  1. Male patients and their female spouses/partners who are of childbearing potential must agree to use a high effective contraception consisting of two forms of birth control detailed in the protocol during the treatment period and for at least 6 days after the dose of the study treatment and refrain from donating sperm during this period
  2. A female patient is eligible if she is not pregnant, not breastfeeding, and at least on of the following conditions applies: (i) not a woman of childbearing potential (WOCBP), (ii) A WOCBP who agrees to follow the contraceptive guidance in the protocol during the treatment period and for at least 6 days after the dose of study treatment and refrain from donating ova during this period
* Patient is capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent and the protocol

Exclusion Criteria:

* Patients who have undergone successful revascularisation on the index leg within 4 weeks of the qualifying event
* Patients with estimated life expectancy <12 months
* Acute limb ischaemia due to thromboembolism within 2 weeks of the qualifying event
* Recent myocardial infarction within 30 calendar days prior to signing informed consent
* Recent stroke within 30 calendar days prior to signing informed consent
* Known history of severe congestive heart failure as determined through review of medical history
* Haemoglobin <8 g/dL, albumin <3 g/dL or other clinically significant abnormalities in the laboratory tests at screening
* Unwilling to complete follow-up evaluation
* Uncontrolled arterial hypertension with systolic blood pressure (SBP) >180 mmHg and/or diastolic blood pressure (DBP) >100 mmHg at screening
* Patients with history of long QT syndrome or whose QTc (calculated according to Bazett formula QTc = QT/ √RR) >470 ms at screening
* Patients with severe left ventricular dysfunction of <40% at screening
* Patients with clinically significant abnormalities in ECG parameters (other than QTc) or in the physical examination at screening that might comprise patient safety
* History of coagulopathy
* Patients having significant renal impairment with estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 as determined by the 4-variable Modification of Diet in Renal Disease (MDRD) equation at Screening, except those patients who are on continuous ambulatory peritoneal dialysis(CAPD) or hemodialysis (HD)
* Significant liver impairment (abnormal Liver Function Tests >3 x upper limit of normal)
* Patients with active Hepatitis B infection (HBsAg positive and HBeAg positive) at screening
* Patient with a positive test for Hepatitis C virus antibody (anti-HCV) at screening
* Patient with known history of infection with human immunodeficiency virus (HIV) or any other active or chronic infection
* Patients with evidence of uncontrolled hypo- or hyperthyroidism
* History active malignancy (as determined through review of medical history), excluding local skin cancer (basal or squamous cell carcinoma)
* Patients unable to provide informed consent
* Known allergy to bovine products
* Receipt of bovine haemoglobin-based oxygen carrier (HBOC) or other HBOC in the past
* Use of an investigational drug or treatment within 12 months prior to signing informed consent; concurrent participation in any other investigational protocol
* Pregnancy and breastfeeding, as well as unwillingness to use effective methods contraception for women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single IV dose of YQ23 - adverse and serious adverse events | From the time of signing informed consent through study completion, a duration of 13 months.
  Incidence of adverse events and serious adverse events
Safety and tolerability of single IV dose of YQ23 - abnormal laboratory values | From the time of signing informed consent through study completion, a duration of 13 months.
  Number of participants with a change in laboratory values of haematology, chemistry or urinalysis which is of clinical significance
Safety and tolerability of single IV dose of YQ23 - 12 lead electrocardiogram (ECG) | From the time of signing informed consent through study completion, a duration of 13 months.
  Number of participants with a change in 12-lead ECG measurements which is of clinical significance
Safety and tolerability of single IV dose of YQ23 - vital signs | From the time of signing informed consent through study completion, a duration of 13 months.
  Number of participants with a change in vital signs of blood pressure, pulse rate, respiratory rate or oral temperature which is of clinical significance
Safety and tolerability of single IV dose of YQ23 - physical examinations | From the time of signing informed consent through study completion, a duration of 13 months.
  Number of participants with a change in physical examination findings which is of clinical significance
Safety and tolerability of single IV dose of YQ23 - major adverse limb events (MALE) | From pre-dose to Month 1
  The incidence of MALE of interest. MALE include amputation (transtibial or above) or any major vascular intervention in the index limb

SECONDARY OUTCOMES:
Efficacy of single dose YQ23 as compared to placebo - all cause mortality | From the time of signing informed consent to Month 12
  Incidence rate of all deaths
Efficacy of single dose YQ23 as compared to placebo - amputation free survival | From pre-dose to Month 12
  Incidence rate of all amputations
Efficacy of single dose YQ23 as compared to placebo - MALE of interest | At month 6 and 12
  Incidence of MALE of interest
Efficacy of single dose YQ23 as compared to placebo - Rutherford classification | From pre-dose, Month 1, 6 and 12
  Change in Rutherford classification
Efficacy of single dose YQ23 as compared to placebo - visual analogue pain scale | From pre-dose, Month 1, 6 and 12
  Change in visual analogue pain scale in a one to ten scale - one reported as no pain while 10 as the most intense pain
Efficacy of single dose YQ23 as compared to placebo - wound healing in size | From pre-dose, Month 1, 6 and 12
  Change in size as measured by length x width x depth in mm
Efficacy of single dose YQ23 as compared to placebo - wound healing by transparent film | From pre-dose, Month 1, 6 and 12
  Change in size as measured by the number of grids in a wound tracing film
Efficacy of single dose YQ23 as compared to placebo - wound healing 100% | From pre-dose, Month 1, 6 and 12
  Number of participants to achieve 100% epithelialization
Efficacy of single dose YQ23 as compared to placebo - wound healing by Wound, Ischemia, and Foot Infection (WIFI) classification system | From pre-dose, Month 1, 6 and 12
  Change in the grading under the WIFI classification system
Efficacy of single dose YQ23 as compared to placebo - transcutaneous oxygen pressure | From pre-dose, 2 hours post-dose, Month 1, 6 and 12
  Change in transcutaneous oxygen pressure (TcPO2)
Efficacy of single dose YQ23 as compared to placebo - quality of life score | From pre-dose, Month 1, 6 and 12
  Change in EuroQol -5 Dimension (EQ-5D) questionnaire
Efficacy of single dose YQ23 as compared to placebo - ankle brachial index (ABI) | From pre-dose, Month 1, 6 and 12
  Change in ABI, a ratio of systolic blood pressure at the ankle to that in the arm
Efficacy of single dose YQ23 as compared to placebo - toe brachial index (TBI) | From pre-dose, Month 1, 6 and 12
  Change in TBI, a ratio of systolic blood pressure at the toe to that in the arm
An optional substudy to assess the pharmacokinetics of YQ23 - maximum observed concentration (Cmax) | From pre-dose, immediately after end of infusion, 0.25, 0.5, 1, 2, 6, 18 (+/-6) and 48 hours post end of infusion
  Plasma level of YQ23 will be serially evaluated following dosing of the study drug to determine the Cmax
An optional substudy to assess the pharmacokinetics of YQ23 - time to Cmax | From pre-dose, immediately after end of infusion, 0.25, 0.5, 1, 2, 6, 18 (+/-6) and 48 hours post end of infusion
  Plasma level of YQ23 will be serially evaluated following dosing of the study drug to determine the time corresponding to occurrence of the Cmax (Tmax)
An optional substudy to assess the pharmacokinetics of YQ23 - Area under the curve (0 to last) | From pre-dose, immediately after end of infusion, 0.25, 0.5, 1, 2, 6, 18 (+/-6) and 48 hours post end of infusion
  Plasma level of YQ23 will be serially evaluated following dosing of the study drug to determine the area under the plasma concentration-time curve (AUC) - AUC from time 0 to the last measurable time point (AUClast)
An optional substudy to assess the pharmacokinetics of YQ23 - Area under the curve (0 to infinity) | From pre-dose, immediately after end of infusion, 0.25, 0.5, 1, 2, 6, 18 (+/-6) and 48 hours post end of infusion
  Plasma level of YQ23 will be serially evaluated following dosing of the study drug to determine the area under the plasma concentration-time curve (AUC) - AUC from time 0 extrapolated to infinity (AUCinf)
An optional substudy to assess the pharmacokinetics of YQ23 - terminal elimination half-life (t1/2) | From pre-dose, immediately after end of infusion, 0.25, 0.5, 1, 2, 6, 18 (+/-6) and 48 hours post end of infusion
  Plasma level of YQ23 will be serially evaluated following dosing of the study drug to determine the t1/2
An optional substudy to assess the pharmacokinetics of YQ23 - total clearance (CL) | From pre-dose, immediately after end of infusion, 0.25, 0.5, 1, 2, 6, 18 (+/- 6) and 48 hours post end of infusion
  Plasma level of YQ23 will be serially evaluated following dosing of the study drug to determine the CL
An optional substudy to assess the pharmacokinetics of YQ23 - volume of distribution during terminal phase (Vz) | From pre-dose, immediately after end of infusion, 0.25, 0.5, 1, 2, 6, 18 (+/- 6) and 48 hours post end of infusion
  Plasma level of YQ23 will be serially evaluated following dosing of the study drug to determine the Vz

CONTACTS AND LOCATIONS:
Overall Officials: Billy Lau, Study Director — New Beta Innovation Limited
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, New Territories
  - Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No